CLINICAL TRIAL: NCT01149720
Title: An Open-Label, Phase 1, Randomized, Two-Treatment, Two-Period, Two-Way Crossover, Relative Bioavailability Study Of A Capsule And A Tablet Formulation Of ARQ 197 In Subjects With Advanced Solid Tumors
Brief Title: Determination of the Relative Bioavailability of ARQ 197 Tablet Formulation With Capsule C Formulation as a Reference in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry); ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARQ197-A-U157
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors
Keywords: Relative bioavailability; ARQ 197
MeSH Terms: interventions — ARQ 197; Capsules; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARQ 197 Capsule, oral (Experimental): Oral BID 360 mg dose (Capsule C: 6 X 60 mg) of ARQ 197 at least 1 hour before or 2 hours after a meal for 7 days
  Interventions: Drug: Tivantinib (ARQ 197) Capsule
- ARQ 197 Tablet, oral (Experimental): Oral BID 360 mg dose (Tablet: 3 x 120 mg) of ARQ 197 under fed conditions for 7 days
  Interventions: Drug: Tivantinib (ARQ 197) Tablet
- ARQ 197 Capsule D, oral (Experimental): Oral BID 360 mg dose (Capsule D: 3 x 120 mg) of ARQ 197 under fed conditions in the extension phase
  Interventions: Drug: Tivantinib (ARQ 197) Capsule D, oral

INTERVENTIONS:
Drug: Tivantinib (ARQ 197) Capsule — Oral BID 360 mg dose (Capsule C: 6 X 60 mg) of ARQ 197 at least 1 hour before or 2 hours after a meal for 7 days
  Other Names: Tivantinib
  Arms: ARQ 197 Capsule, oral
Drug: Tivantinib (ARQ 197) Tablet — Oral BID 360 mg dose (Tablet: 3 x 120 mg) of ARQ 197 under fed conditions for 7 days
  Other Names: Tivantinib
  Arms: ARQ 197 Tablet, oral
Drug: Tivantinib (ARQ 197) Capsule D, oral — Oral BID 360 mg dose (Capsule D: 3 x 120 mg) of ARQ 197 under fed conditions in the extension phase
  Other Names: Tivantinib
  Arms: ARQ 197 Capsule D, oral

SUMMARY:
This is a Phase 1, randomized, open label, 2 treatment, 2 period, 2-way crossover study, with an extension phase design in which the steady state PK of ARQ 197 will be investigated using the tablet administered in fed state (test treatment) and capsule administered at least 1 hour before or 2 hours after a meal (reference treatment) in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically or cytologically confirmed advanced solid tumor at screening.
* Male or female equal or greater than 18 years of age.
* All female subjects of childbearing potential must each have a negative serum pregnancy test result before initiating study treatment.
* An Eastern Cooperative Oncology Group (ECOG) performance status equal or less than 2
* Adequate bone marrow, liver, and renal function, defined as:

  * Platelet count equal or greater than 75 x 10(9)/L
  * Hemoglobin (Hb) equal or greater than 9.0 g/dL
  * Absolute neutrophil count (ANC) equal or greater than 1.5 x 10(9)/L
  * Total bilirubin equal or less than 1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) equal or less than 3 x ULN (equal or less than 5 x ULN for subjects with liver metastases)
  * Serum creatinine equal or less than 1.5 x ULN

Exclusion Criteria:

* History of cardiac disease: Active coronary artery disease (CAD), defined as myocardial infarction (MI), unstable angina, coronary bypass graft (CABG), or stenting within 6 months prior to study entry (an MI that occurred > 6 months prior to study entry is permitted)
* Evidence of uncontrolled bradycardia or other cardiac arrhythmia defined as equal or greater than Grade 2 according to NCI CTCAE, version 4.0, or uncontrolled hypertension
* Active, clinically serious infection(s) defined as equal or greater than Grade 2 according to NCI CTCAE, version 4.0.
* Known metastatic brain or meningeal tumors, unless the subject is > 3 months from definitive therapy and clinically stable (supportive therapy with steroids or anticonvulsant medications is allowed) with respect to the tumor at the time of first dose of study drug.
* Prior therapy with mesenchymal-epithelial transition factor (c-MET) inhibitors, including ARQ 197.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Determination of the relative bioavailability of ARQ 197 tablet formulation with capsule C formulation | 14 days
  The primary endpoints are the area under the concentration time curve from time of dosing until 12 hours post-dose (AUC0-12) and maximum observed concentration in plasma (Cmax) of ARQ 197 following the administration of the tablet (fed conditions) and capsule formulation (at least 1 hour before or 2 hours after a meal).

SECONDARY OUTCOMES:
Assessment of additional pharmacokinetic parameters of ARQ 197 tablet formulation and capsule C formulation | 14 days
  Time until Cmax (tmax), apparent oral clearance (CL/F), and apparent volume of distribution (V/F) of ARQ 197, and if possible, minimum observed concentration (Cmin) and average observed concentration (Cavg) following the administration of the tablet (fed conditions) and capsule formulation (at least 1 hour before or 2 hours after a meal)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Premiere Oncology, Santa Monica, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/